CLINICAL TRIAL: NCT04709848
Title: Seroprevalence and Impact of Screening for Strongyloides Stercoralis in Bone Marrow Transplant Recipients in the UK
Brief Title: Strongyloides Stercoralis in Bone Marrow Transplant Recipients in the UK
Acronym: SSSSBMTUK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH6406
Record Dates: First submitted 2021-01-05; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Strongyloidiasis; Bone Marrow Transplant Infection
MeSH Terms: conditions — Strongyloidiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-screening group: Individuals undergoing bone marrow transplantation Jun 2018 - July 2020
  Interventions: Other: None - standard of care
- Screened group: Individuals undergoing bone marrow transplantation July 2020 - July 2021
  Interventions: Other: None - standard of care

INTERVENTIONS:
Other: None - standard of care — Observational study only. Pre-screening group were not screened for Strongyloides, as per the standard of care at the time. Screened group were screened for Strongyloides, because the standard of care at our centre changed.

SUMMARY:
Strongyloidiasis is a worm infection which affects more than 100 million people, mostly in Africa, Asia and Latin America, and can cause severe illness in people with reduced immunity. In the UK, the number of people with Strongyloides is not known.

At Imperial College Healthcare NHS Trust (ICHNT) , screening for Stongyloides has recently been introduced as a standard-of-care for all patients undergoing BMT.

In this study, investigators will perform two cross-sectional surveys and report the prevalence of Strongyloides in BMT recipients at ICHNT , as well as comparing clinical outcomes before/after the introduction of routine testing.

DETAILED DESCRIPTION:
Strongyloidiasis is a worm infection which affects more than 100 million people, mostly in Africa, Asia and Latin America. Infection can persist for decades, and usually causes mild symptoms. In some people with reduced immune systems (for example those who have bone marrow transplantation), the worms can multiply and cause severe illness and death.

In the UK, the number of people with Strongyloides is not known. However, in many other non-tropical countries, rates are high in immigrant populations (including those who are having bone marrow transplantation, BMT).

At ICHNT, screening for Stongyloides has recently been introduced as a standard-of-care for all patients undergoing BMT. All adult patients with forthcoming BMT at ICHNT will now be screened. Additionally, any patients who have already undergone BMT in the last two years will be screened as part of a look-back exercise as part of their clinical care.

In this study, investigators will perform two cross-sectional surveys. Those who underwent BMT between Jun 2018 - July 2020 will form a 'pre-screening group', and those between July 2020 - July 2021 will form a 'screened group'. It is anticipated that 320 participants will be included in the pre-screening group and 160 in the screened-group (total 480).

Data will be collected retrospectively and the prevalence of Strongyloides in BMT recipients at ICHNT will be reported. Comparison of clinical outcomes between the first and second groups will be undertaken, in order to determine whether the introduction of screening has had an impact.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Under care of Haematology at ICHNT
* Undergoing BMT Jun 2018 - July 2020 ('pre-screening group') or July 2020 - July 2021 ('screened group')

Exclusion Criteria:

* Age < 18 years (i.e. managed as paediatric BMT)
* Previous BMT but no Strongyloides serology result available at the time of data collection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals under the care of Haematology at ICHNT
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Strongyloides seropositivity | Baseline

SECONDARY OUTCOMES:
BMT outcome | Within first 12 months after BMT
  Bloodstream infection
BMT outcome | Within first 12 months after BMT
  Respiratory disease
BMT outcome | Within first 12 months after BMT
  Clinically significant diarrhoea
BMT outcome | Within first 12 months after BMT
  CNS infection
BMT outcome | Within first 12 months after BMT
  Graft vs. host disease
BMT outcome | Within first 12 months after BMT
  Length-of-hospital-stay
BMT outcome | Within first 12 months after BMT
  Antibiotic usage (defined daily doses)
BMT outcome | Within first 12 months after BMT
  ICU admission
BMT outcome | Within first 12 months after BMT
  Strongyloides hyperinfection syndrome
BMT outcome | Within first 12 months after BMT
  Mortality

IPD SHARING:
Plan to Share IPD: No